CLINICAL TRIAL: NCT03278028
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study of A-101 Topical Solution Applied Twice a Week in Subjects With Common Warts
Brief Title: A Study of A-101 Topical Solution Administered Twice a Week in Subjects With Common Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-101-WART-203
Record Dates: First submitted 2017-08-18; First posted 2017-09-11 (Actual); Results first posted 2019-03-29 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Common Wart
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): A-101 Topical Solutions
  Interventions: Drug: A-101 Topical Solution
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: A-101 Vehicle Solution

INTERVENTIONS:
Drug: A-101 Topical Solution — A-101 Topical Solution
  Arms: Active
Drug: A-101 Vehicle Solution — A-101 Vehicle Solution
  Arms: Vehicle

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of A-101 compared to Vehicle when applied to 1 Target common wart on the trunk or extremities twice a week.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effectiveness of A-101 compared to Vehicle when applied to 1 Target common wart on the trunk or extremities twice a week.

The secondary objectives of this study are to evaluate the clinical effect of A-101 when applied to all treated Warts (Target Warts plus Non-Target Warts) twice a week, duration of response in all treated Warts (Target Warts plus Non-Target Warts), and safety of A-101.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to comprehend and is willing to sign an informed consent/assent for participation in this study.
* Male or female ≥ 8 years old.
* Subject chemistry and complete blood count results are within normal limits. If any of the laboratory values are outside normal range, the treating investigator must assess the value/s as NOT clinically significant and document this in the subject's medical chart in order for the subject to be eligible for randomization.
* Woman of childbearing potential (WOCBP) must have a negative urine pregnancy test within 14 days of the first application of study drug and agree to use an active method of birth control for the duration of the study.
* Subject is non-pregnant and non-lactating.
* Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair the evaluation of any Target and Non-Target Warts or which exposes the subject to an unacceptable risk by study participation.
* Subject is willing and able to follow all study instructions and to attend all study visits.

Exclusion Criteria:

* Subject has clinically atypical warts on the trunk or extremities.
* Subject is immunocompromised (e.g., due to chemotherapy, systemic steroids, genetic immunodeficiency, transplant status, etc.)
* Subject has a history of Human Immunodeficiency Virus (HIV) infection
* Subject has had any Human Papilloma Virus (HPV) vaccine within 1 year prior to Visit 1
* Subject has a history of sensitivity to any of the ingredients in the study medications.
* Subject has any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage), or condition (e.g., sunburn, excessive hair, open wounds) that, in the opinion of the investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations.
* Participation in another therapeutic investigational drug trial in which administration of an investigational study medication occurred with 30 days prior to Visit 1.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Shanler, MD, Study Director — Aclaris Therapeutics
Locations (16):
- United States (16):
  - Aclaris Investigational Site, Glendale, Arizona
  - Aclaris Investigational Site, Fort Smith, Arkansas
  - Aclaris Investigational Site, Encinitas, California
  - Aclaris Investigational Site, Los Angeles, California
  - Aclaris Investigational Site, Denver, Colorado
  - Aclaris Investigational Site, Omaha, Nebraska
  - Aclaris Investigational Site, Albuquerque, New Mexico
  - Aclaris Investigational Site, Rochester, New York
  - Aclaris Investigational Site, High Point, South Carolina
  - Aclaris Investigational Site, Knoxville, Tennessee
  - Aclaris Investigational Site, Nashville, Tennessee
  - Aclaris Investigational Site, College Station, Texas
  - Aclaris Investigational Site, Houston, Texas
  - Aclaris Investigational Site, Salt Lake City, Utah
  - Aclaris Investigational Site, Lynchburg, Virginia
  - Aclaris Investigational Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Vehicle
Started | 81 | 78
Completed | 77 | 76
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active: A-101 Topical Solution
  A-101 Topical Solution: A-101 Topical Solution
- Total: Total of all reporting groups
Arm/Group | Active | Vehicle | Total
Number analyzed (Participants) | 81 | 78 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.96 (18.09) | 41.56 (17.42) | 39.73 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 43 | 91
  Male | 33 | 35 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 16 | 29
  Not Hispanic or Latino | 65 | 55 | 120
  Unknown or Not Reported | 3 | 7 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 1 | 4 | 5
  White | 78 | 70 | 148
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 81 | 78 | 159

OUTCOME MEASURES:

1. Primary Outcome: Physician's Wart Assessment
Description: Physician's Wart Assessment Grade Descriptor 0 Clear: No visible wart. No further treatment is indicated.
  1. Near Clear: A visible wart that is less than 3 mm in maximal diameter (or length)
  2. A visible wart ≥ 3 mm and < 6 mm in maximal diameter (or length)
  3. A visible wart ≥ 6 mm in maximal diameter (or length)
Time Frame: Day 57
Population: Per-Protocol (PP)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Vehicle
Number analyzed (Participants) | 79 | 78
score on a scale | 1.52 (1.06) | 2.23 (0.66)

ADVERSE EVENTS:
Time Frame: 78 days; Treatment-emergent adverse events (TEAEs) had a start date on or after the date of Visit 2 (study day 1) and treatment-emergent serious adverse events had a start date on or after the date of Visit 1 (Screening). Collection continued through visit 11 (Day 78)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation subject administered a study medication(s) and that did not necessarily have a causal relationship with the study medication.
  Safety summaries by study medication group will include listings by study medication of adverse events incidences within each MedDRA System Organ Class, and changes from pre-application values in vital signs.
Arm/Group | Active | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/78
Other Adverse Events (participants affected / at risk) | 28/81 | 19/78
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=81) | Vehicle (N=78)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application Site Pain (General disorders) | 1 (1) | 0 (0)
Food Allergy (Immune system disorders) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 1 (1) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1)
Eye Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Localised Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post Operative Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0)
Liver Function Test Increased (Investigations) | 1 (1) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Squamous Cell Carcinoma of Head and Neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Device Dislocation (Product Issues) | 0 (0) | 1 (1)
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Haemorrage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03278028/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03278028/SAP_001.pdf